CLINICAL TRIAL: NCT04450576
Title: HbA1c as an Early Serologic Marker for the Hemodynamic Progression of Stage A Heart
Brief Title: HbA1c as an Early Serologic Marker for the Hemodynamic Progression of Stage A Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Parkview Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PIRB74
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Glycosylated hemoglobin — Glycosylated hemoglobin levels associated with correlative measures of diastolic cardiac function
  Other Names: Echocardiogram

SUMMARY:
In a retrospective community based cohort study from Pueblo County Colorado which has a higher population proportion of metabolic syndrome and diabetes mellitus, we hope to clarify and quantify an association of the AGE HBa1c elevation with the early subclinical hemodynamic changes of diabetic cardiomyopathy as measured by LAV, LVM, E/A ratio, E/e' ratio and BNP in patients with stage A heart failure.

DETAILED DESCRIPTION:
The classic association of glycemic control, as represented by HBa1c, with progression or improvement of microvascular and macrovascular clinical complications has been well documented. Additionally, while the association of HBa1c elevation with a syndrome described as diabetic cardiomyopathy has also been well documented, the use of the advanced glycation end product axis (AGE/sRAGE/esRAGE which includes HBa1c) as markers for the early subclinical hemodynamic changes of diabetic cardiomyopathy has been suggested but less well characterized or utilized. Stage A heart failure is defined as persons with normal cardiac structure and function who have predisposing subclinical risks for cardiovascular disease. Estimates suggest that Stage A heart failure may comprise up to 56% of any community's patient population and are patients most commonly seen in non-specialty primary care clinics. In light of newer cardiometabolic agents which show promise in cardiovascular disease primary prevention, these patients may be an important target for preventative cardiometabolic care. In a retrospective community based cohort study from Pueblo County Colorado which has a higher population proportion of metabolic syndrome and diabetes mellitus, we hope to clarify and quantify an association of the AGE HBa1c elevation with the early subclinical hemodynamic changes of diabetic cardiomyopathy as measured by LAV, LVM, E/A ratio, E/e' ratio and BNP in patients with stage A heart failure.

Methods: Retrospective cohort analysis by chart review of patients presenting to Parkview Medical Center's inpatient service and outpatient clinics who obtained a full resting echo characterized by normal cardiac structure and function in conjunction with HBa1c and BNP levels within a 3 month time window. Using multiple regression analysis of the dependent variables LAV, LVM, E/A ratio, E/e' ratio and BNP, powered to detect a 5% change in LAV in conjunction with rising HBa1c levels characterized as normal (<5.7), metabolic syndrome (5.7-6.4) or diabetic (>6.4) after controlling for the presence of hypertension and coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Stage A heart failure on basis of metabolic criteria

Exclusion Criteria:

* LV dysfunction, valvular heart disease, hypertension and CAD

Age Groups: Child, Adult, Older Adult
Study Population: Stage A heart failure patients who have had a Glycosylated hemoglobin, BNP and Echocardiogram with any 3 month contiguous time period during the lookback period
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Left Atrial volume | 3 months
  Echocardiogram

SECONDARY OUTCOMES:
BNP | 3 months
  Serum total values in pg/ml
E/e' | 3 months
  Echocardiogram measure of the ratio of early LA to LV diastolic inflow velocity (E) to tissue doppler measure of mitral annular early diastolic velocity (e') in m/sec. This is a marker of left atrial pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Duffee, MD, Principal Investigator — Parkview Medical Center
Locations (1):
- Parkview Medical Center, Pueblo, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
no plan to make IPD available outside our facility

REFERENCES:
- [Background] Fowler MJ. Microvascular and macrovascular complications of diabetes. Clinical Diabetes. 2011;29(3):116-122.
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Beckman JA, Creager MA, Libby P. Diabetes and atherosclerosis: epidemiology, pathophysiology, and management. JAMA. 2002 May 15;287(19):2570-81. doi: 10.1001/jama.287.19.2570. PMID 12020339
- [Background] Fox CS, Coady S, Sorlie PD, Levy D, Meigs JB, D'Agostino RB Sr, Wilson PW, Savage PJ. Trends in cardiovascular complications of diabetes. JAMA. 2004 Nov 24;292(20):2495-9. doi: 10.1001/jama.292.20.2495. PMID 15562129
- [Background] van Heerebeek L, Hamdani N, Handoko ML, Falcao-Pires I, Musters RJ, Kupreishvili K, Ijsselmuiden AJ, Schalkwijk CG, Bronzwaer JG, Diamant M, Borbely A, van der Velden J, Stienen GJ, Laarman GJ, Niessen HW, Paulus WJ. Diastolic stiffness of the failing diabetic heart: importance of fibrosis, advanced glycation end products, and myocyte resting tension. Circulation. 2008 Jan 1;117(1):43-51. doi: 10.1161/CIRCULATIONAHA.107.728550. Epub 2007 Dec 10. PMID 18071071
- [Background] Levelt E, Gulsin G, Neubauer S, McCann GP. MECHANISMS IN ENDOCRINOLOGY: Diabetic cardiomyopathy: pathophysiology and potential metabolic interventions state of the art review. Eur J Endocrinol. 2018 Apr;178(4):R127-R139. doi: 10.1530/EJE-17-0724. Epub 2018 Feb 12. PMID 29440374
- [Background] Singh VP, Bali A, Singh N, Jaggi AS. Advanced glycation end products and diabetic complications. Korean J Physiol Pharmacol. 2014 Feb;18(1):1-14. doi: 10.4196/kjpp.2014.18.1.1. Epub 2014 Feb 13. PMID 24634591
- [Background] Jia G, DeMarco VG, Sowers JR. Insulin resistance and hyperinsulinaemia in diabetic cardiomyopathy. Nat Rev Endocrinol. 2016 Mar;12(3):144-53. doi: 10.1038/nrendo.2015.216. Epub 2015 Dec 18. PMID 26678809
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202
- [Background] Ammar KA, Jacobsen SJ, Mahoney DW, Kors JA, Redfield MM, Burnett JC Jr, Rodeheffer RJ. Prevalence and prognostic significance of heart failure stages: application of the American College of Cardiology/American Heart Association heart failure staging criteria in the community. Circulation. 2007 Mar 27;115(12):1563-70. doi: 10.1161/CIRCULATIONAHA.106.666818. Epub 2007 Mar 12. PMID 17353436
- [Background] Mahaffey KW, Jardine MJ, Bompoint S, Cannon CP, Neal B, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Capuano G, de Zeeuw D, Greene T, Levin A, Pollock C, Sun T, Wheeler DC, Yavin Y, Zhang H, Zinman B, Rosenthal N, Brenner BM, Perkovic V. Canagliflozin and Cardiovascular and Renal Outcomes in Type 2 Diabetes Mellitus and Chronic Kidney Disease in Primary and Secondary Cardiovascular Prevention Groups. Circulation. 2019 Aug 27;140(9):739-750. doi: 10.1161/CIRCULATIONAHA.119.042007. Epub 2019 Jul 11. PMID 31291786
- [Background] From AM, Scott CG, Chen HH. The development of heart failure in patients with diabetes mellitus and pre-clinical diastolic dysfunction a population-based study. J Am Coll Cardiol. 2010 Jan 26;55(4):300-5. doi: 10.1016/j.jacc.2009.12.003. PMID 20117433
- [Background] Pueblo County 2016 Community Health Status report.